CLINICAL TRIAL: NCT03691077
Title: A Prospective Study Evaluating the Effect of Ocrelizumab on Brain Innate Immune Microglial Cells Activation in Multiple Sclerosis Using PET-MRI With 18F-DPA714
Brief Title: Effect of Ocrelizumab on Brain Innate Immune Microglial Cells Activation in MS Using PET-MRI With 18F-DPA714
Acronym: INN-MS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Roche Pharma AG (Industry); Institut du Cerveau et de la Moelle épinière (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P170702J
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Relapse; Primary Progressive Multiple Sclerosis
Keywords: Multiple Sclerosis; Ocrelizumab; Microglial cells Activation; PET-IRM; 18F-DPA714
MeSH Terms: conditions — Multiple Sclerosis; Recurrence; Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab

STUDY DESIGN:
Intervention Model Description: The first dose of ocrelizumab will be administered as two 300-mg IV infusions (600 mg total) in 250 mL 0.9% sodium chloride each separated by 14 days (i.e., Days 1 and 15), followed by one 600-mg IV infusion in 500 mL 0.9% sodium chloride every subsequent doses (i.e., every 24 weeks) for 72 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocrelizumab (Experimental): The first dose of ocrelizumab will be administered as two 300-mg IV infusions (600 mg total) in 250 mL 0.9% sodium chloride each separated by 14 days (i.e., Days 1 and 15), followed by one 600-mg IV infusion in 500 mL 0.9% sodium chloride every subsequent doses (i.e., every 24 weeks) for 72 weeks.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — The first dose of ocrelizumab will be administered as two 300-mg IV infusions (600 mg total) in 250 mL 0.9% sodium chloride each separated by 14 days (i.e., Days 1 and 15), followed by one 600-mg IV infusion in 500 mL 0.9% sodium chloride every subsequent doses (i.e., every 24 weeks) for 72 weeks.

SUMMARY:
Ocrelizumab is a humanized anti-CD20 monoclonal antibody that showed in phase III trials a powerful effect on relapse rate and lesion load accumulation in the relapsing form of multiple sclerosis (RMS). This therapeutic agent also showed for the first time a significant reduction of disability progression in Primary Progressive Multiple Sclerosis (PPMS) patients, whereas all other anti-inflammatory drugs had failed to do so in well-conducted studies. This raises the possibility that ocrelizumab, beyond its effects on the adaptive immune system activation underlying white matter lesions and clinical relapses, could beneficially influence other mechanisms involved in the progressive phase of the disease, such as the innate immune microglial cells activation, that has been described to persist in a diffuse manner in the Central Nervous system (CNS). To date the activation of these cells is not accessible to classical Magnetic Resonance Imaging (MRI) techniques, impeding the full investigation of the therapeutic efficacy of drugs such as ocrelizumab.

DETAILED DESCRIPTION:
The first dose of ocrelizumab will be administered as two 300-mg IV infusions (600 mg total) in 250 mL 0.9% sodium chloride each separated by 14 days (i.e., Days 1 and 15), followed by one 600-mg IV infusion in 500 mL 0.9% sodium chloride every subsequent doses (i.e., every 24 weeks) for 72 weeks.

Premedication with 100 mg of methylprednisolone (or an equivalent) approximately 30 minutes prior to each ocrelizumab infusion and additional premedication with an antihistaminic drug (e.g., diphenhydramine) approximately 30 - 60 minutes before each infusion of ocrelizumab to reduce the frequency and severity of infusion-related reactions (IRRs). The addition of an antipyretic (e.g., acetaminophen/ paracetamol) may also be considered.

Patients will undergo PET scan with 18F-DPA714 and MRI exams at different time points as mentioned in the assessment table.

Disease will be clinically monitored at different time points with classical tests including EDSS, MSFC, BICAMS.

Laboratory analyses on complete blood count, lymphocytes subsets count, neurofilament will be done. Analyses will not be limited to the above mentioned list.

Pregnancy tests and genetics will be done. An optional lumbar puncture will be performed at baseline to assess cytokinic profile predictive of disease evolution and cortical pathology. Patients who refuse to have a lumbar puncture can be included in the clinical trial if they have eligibility criteria.

TSPO polymorphism will be checked at baseline with other screening lab tests.

ELIGIBILITY:
Inclusion criteria for all MS subgroups:

1. Signed informed consent form
2. Able to comply with the study protocol, in the investigator's judgment
3. Social security registration
4. Age 18 - 60 years, inclusive
5. For women of childbearing potential: agreement to use an acceptable birth control method during the treatment period and for at least 12 months after the last dose of study drug.

RMS

1. Have a definite diagnosis of RMS, confirmed as per the revised McDonald 2010 criteria (Polman et al. 2011);
2. Absence of history of Secondary Progressive Multiple Sclerosis (SPMS) or history of Primary Progressive Multiple Sclerosis (PPMS)
3. Have an active disease: Activity determined by clinical relapses and/or MRI activity (contrast-enhancing lesions; new or unequivocally enlarging T2 lesions assessed at least annually (Lublin et al. 2014))
4. Neurological stability for ≥30 days prior to both screening and baseline
5. EDSS of 0.0 to 5.5, inclusive, at screening
6. Have a length of disease duration, from first symptom, of < 15 years
7. Have received no more than first line injectable treatments (i.e. IFNs and GA, possible switchs within this class) + 1 other treatment (e.g. teriflunomide, DMF, fingolimod, natalizumab, no switch allowed within this group). More details in section 6.1.1.2.1
8. Have a suboptimal response to the last received DMT: a suboptimal response is defined by having at least one of the following events while being on a stable dose of the same DMT for at least 6 months:

   1. One or more clinically reported relapse(s)
   2. OR one or more T1 Gd-enhanced lesion(s)
   3. OR one or more new and/or enlarging T2 lesions on MRI
9. In addition, in patients receiving stable doses of the same approved DMT for more than a year, at least one of the above events must have occurred within the last 12 months of treatment with this DMT.

RMS

1. Diagnosis of SPMS according to Lublin et al. 2014 criteria
2. Prior history of RRMS (Have a definite diagnosis of RRMS, confirmed as per the revised McDonald 2010 criteria
3. Have an active disease during the two years preceding the study entry: Activity determined by clinical relapses and/or MRI activity (contrast-enhancing lesions; new or unequivocally enlarging T2 lesions assessed at least annually (Lublin et al. 2014))
4. Evidence of any disability progression unrelated to relapse within the 2 year period prior to study baseline. Progression in the last year will be reported by the treating physician and documented using a disease progression rating system checklist (see Appendix 1)
5. Progression is defined as steadily increasing objectively documented neurologic dysfunction/disability without unequivocal recovery (fluctuations and phases of stability may occur) (Lublin, 2014)
6. Absence of history of Primary Progressive Multiple Sclerosis or Progressive Relapsing Multiple Sclerosis at screening
7. EDSS at screening ≤ 6.5points
8. Score of ≥ 2.0 on the Functional Systems (FS) scale for the pyramidal system that is due to lower extremity findings
9. Disease duration from the onset of Secondary Progressive MS symptoms of less than 10 years if baseline EDSS ≤5
10. Disease duration from the onset of Secondary Progressive MS symptoms of less than 15 years if baseline EDSS >5
11. Have received no more than first line treatments (either injectable, i.e. IFNs and GA, or oral, either teriflunomide and dimethyl fumarate, possible switchs within this group) + 1 second line treatment (e.g., fingolimod, natalizumab, no switch allowed within this group).

PPMS

1. Diagnosis of PPMS in accordance with the 2010 revised McDonald criteria :
2. One year of disease progression (retrospectively or prospectively determined)
3. Plus 2 of the 3 following criteria :

   1. Evidence for DIS in the brain based on ≥ 1 T2 lesions in at least 1 area characteristic for MS (periventricular, juxtacortical, or infratentorial)
   2. Evidence for DIS in the spinal cord based on ≥ 2 T2 lesions in the cord
   3. Positive CSF (isoelectric focusing evidence of oligoclonal bands and/or elevated IgG index)
4. Absence of history of Relapsing Remitting Multiple Sclerosis, Secondary Progressive, or Progressive Relapsing Multiple Sclerosis at screening
5. Evidence of any disability progression unrelated to relapse within the 2 year period prior to study baseline. Progression in the last 2 year will be reported by the treating physician and documented using a disease progression rating system checklist (see Appendix 1)
6. EDSS at screening between 2.0 and 6.5 points
7. Score of ≥ 2.0 on the Functional Systems (FS) scale for the pyramidal system that is due to lower extremity findings
8. Disease duration from the onset of MS symptoms of less than 10 years if baseline EDSS ≤5
9. Disease duration from the onset of MS symptoms of less than 15 years if baseline EDSS >5

Healthy volunteers (20 subjects):

1. Signed informed consent form
2. Able to comply with the study protocol, in the investigator's judgment
3. Social security registration
4. Age 18 - 60 years, inclusive
5. For women of childbearing potential: agreement to use an acceptable birth control method during the research period and for at least 1 cycle after the PET-MRI.

   1. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
   2. The following are acceptable contraceptive methods: progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action, male or female condom with or without spermicide, and cap, diaphragm, or sponge with spermicide. A combination of male condom with cap, diaphragm, or sponge with spermicide (double barrier methods) is considered acceptable
   3. Pregnancy tests will be performed at each study visit for women of childbearing potential.

Exclusion Criteria:

1. Inability to complete an MRI (contraindications for MRI include but are not restricted to weight ≥ 140 kg, pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, contraindication to gadoteric acid etc.).
2. Impossibility to complete a PET scan: pregnancy, nuclear medicine irradiation in the year preceding baseline visit for clinical research and one year after the end of their participation in the study, lactation.
3. Known presence of other neurological disorders, including but not limited to, the following:

   1. History of ischemic cerebrovascular disorders (e.g., stroke, transient ischemic attack) or ischemia of the spinal cord
   2. History or known presence of CNS or spinal cord tumor (e.g., meningioma, glioma)
   3. History or known presence of potential metabolic causes of myelopathy (e.g., untreated vitamin B12 deficiency)
   4. History or known presence of infectious causes of myelopathy (e.g., syphilis, Lyme disease, human T-lymphotropic virus 1 (HTLV-1), herpes zoster myelopathy)
   5. History of genetically inherited progressive CNS degenerative disorder (e.g., hereditary paraparesis; MELAS [mitochondrial myopathy, encephalopathy, lactic acidosis, stroke] syndrome)
   6. Neuromyelitis optica
   7. History or known presence of systemic autoimmune disorders potentially causing progressive neurologic disease (e.g., lupus, anti-phospholipid antibody syndrome, Sjogren's syndrome, Behçet's disease)
   8. History or known presence of sarcoidosis
   9. History of severe, clinically significant brain or spinal cord trauma (e.g., cerebral contusion, spinal cord compression) - General Health:

1. Pregnancy or lactation 2. Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressant drugs during the course of the study 3. History or currently active primary or secondary immunodeficiency 4. Lack of peripheral venous access 5. Significant, uncontrolled disease, such as cardiovascular (including cardiac arrhythmia), pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine or gastrointestinal or any other significant disease that may preclude patient from participating in the study 6. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies 7. Congestive heart failure (New York Heart Association [NYHA] III or IV functional severity) 8. Known active bacterial, viral, fungal, mycobacterial infection or other infection [including tuberculosis [TB] or atypical mycobacterial disease (but excluding fungal infection of nail beds)] or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks prior to baseline visit or oral antibiotics within 2 weeks prior to baseline visit; Note: Active infections should be treated and effectively controlled before possible inclusion in the study 9. History or known presence of recurrent or chronic infection 10. History of malignancy, including solid tumors and hematological malignancies, except basal cell carcinoma, in situ squamous cell carcinoma of the skin, and in situ carcinoma of the cervix of the uterus that have been previously completely excised with documented, clear margins 11. History of alcohol or drug abuse within 24 weeks prior to baseline 12. History or laboratory evidence of coagulation disorders 13. History of major opportunistic infections (i.e. cryptococcosis, Pneumocystis pneumonia, progressive multifocal leukoencephalopathy [PML]) 14. History of recurrent aspiration pneumonia requiring antibiotic therapy 15. Hypersensitivity to the active substance or to any of the excipients (Sodium Acetate Trihydrate, Glacial Acetic Acid, Trehalose Dihydrate, Polysorbate 20, Water for Injection)

* Laboratory Findings:

  1. TSPO polymorphism indicating a low affinity profile.
  2. Positive serum β human chorionic gonadotropin (hCG) measured at screening and before each PET-Scan procedure
  3. Positive screening tests for hepatitis B (hepatitis B surface antigen [HBsAg] positive, or positive hepatitis B core antibody [total HBcAb] confirmed by a positive viral DNA polymerase chain reaction [PCR]) or hepatitis C (HepCAb)
  4. Lymphocyte count below lower limit of normal (LLN)
  5. CD4 count <300/μL.
  6. Absolute neutrophil count <1.0 × 103/µL
* Medications:

  1. Receipt of a live vaccine or attenuated live vaccine within 6 weeks prior to the baseline visit. In rare cases when patient requires vaccination with a live vaccine, the screening period may be extended but cannot exceed 8 weeks
  2. Treatment with any investigational agent within 24 weeks of screening or five half-lives of the investigational drug (whichever is longer) or treatment with any experimental procedures for MS (e.g., treatment for chronic cerebrospinal venous insufficiency)
  3. Treatment with Flumitrazepam, triazolam, diazepam
* Treatment of Multiple Sclerosis:

  1. Previous treatment with B-cell targeted therapies (i.e., rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab)
  2. Systemic corticosteroid therapy within 4 weeks prior to screeningii
  3. Treatment with IV immunoglobulin (Ig) within 12 weeks prior to baseline
  4. Any previous treatment with alemtuzumab, daclizumab, anti-CD4, total body irradiation or bone marrow transplantation
  5. Any previous treatment with biotin in the last month prior to screening
  6. Previous treatment with mitoxantrone, cyclosporine or cladribine in the last 96 weeks
  7. Previous treatment with azathioprine, cyclophosphamide, mycophenolate mofetil,methotrexate, or laquinimod in the last 24 weeks
  8. Previous treatment with teriflunomide, unless an accelerated elimination procedure is implemented before screening visit. Accelerated elimination procedure after stopping treatment with teriflunomide:

     1. cholestyramine 8g is administered 3 times daily for a period of 11 days, or cholestyramine 4g three times a day can be used, if cholestyramine 8g three times a day is not well tolerated,
     2. alternatively, 50g of activated powdered charcoal is administered every 12 hours for a period of 11 days
  9. Previous treatment with natalizumab in the last 12 weeks
  10. Previous treatment with fingolimod or dimethyl fumarate if at baseline the lymphocyte count is below lower limit of normality (LLN). Apart from the lymphocytes count within normal ranges, 12 weeks of a washout period of fingolimod or dimethylfumarate would be required before the start of ocrelizumab administration
  11. History of recurrent aspiration pneumonia requiring antibiotic therapy
  12. Treatment with fampridine/dalfamipridine (Fampyra®)/Ampyra®) unless on stable dose for ≥ 30 days prior to screening. Wherever possible, patients should remain on stable doses throughout the 96-week treatment period
  13. Treatment with β interferons, glatiramer acetate, plasmapheresis, or other immunomodulatory therapies within 4 weeks prior to baselinei

Healthy volunteers:

1. Inability to complete an MRI (contraindications for MRI include but are not restricted to weight ≥ 140 kg, pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, contraindication to acid gadoteric etc.)
2. Impossibility to complete a PET scan: pregnancy, nuclear medicine irradiation in the year preceding baseline visit for clinical research
3. Known presence of any neurological disorders
4. Pregnancy or lactation
5. Lack of peripheral venous access
6. Significant, uncontrolled disease, such as cardiovascular (including cardiac arrhythmia), pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine or gastrointestinal infectious, neoplasic or any other significant disease that may preclude patient from participating in the study
7. History of alcohol or drug abuse within 24 weeks prior to baseline
8. TSPO polymorphism indicating a low affinity profile.
9. Treatment with Flumitrazepam, triazolam, diazepam

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Determine if ocrelizumab treatment is associated with a decrease in the extent of brain white matter microglial activation. | from baseline to month 24
  Percent change in the extent of 18FDPA714 positive voxels in the total white matter from baseline to month 24 in the whole cohort of MS patients.

SECONDARY OUTCOMES:
Decrease of microglial activation as measured by [18F]DPA-714 PET in normal appearing white matter | between baseline and months 6 and 24
  Percent change in extent of 18FDPA714 positive voxels in normal appearing white matter between baseline and months 6 (short-term) and 24 (long-term) in the whole cohort, in RMS cohort (global and splitted in RRMS and RMS having reached the SPMS phase) and in PPMS cohort
decrease of microglial activation as measured by [18F]DPA-714 PET in the total white matter | from baseline to months 24
  Percent change in extent of [18F]-DPA-714 positive voxels in the total white matter from baseline to month 24, in PPMS cohort and in RMS cohort (whole cohort and subgroups of RRMS and SPMS patients).
decrease of microglial activation as measured by [18F]DPA-714 PET in white matter lesions | between baseline and months 6 and 24
  Percent change in extent of 18FDPA714 positive voxels in white matter lesions between baseline to months 6 and 24, in the whole cohort, in RMS cohort (global and splitted in RRMS and RMS having reached the SPMS phase) and in PPMS cohort.
decrease of microglial activation as measured by [18F]DPA-714 PET in white matter perilesional areas | between baseline to months 6 and 24
  Percent change in extent of 18FDPA714 positive voxels in white matter perilesional areas between baseline to months 6 and 24 in the whole cohort, in RMS cohort (global and splitted in RRMS and RMS having reached the SPMS phase) and in PPMS cohort.
decrease of microglial activation as measured by [18F]DPA-714 PET in in number of plaques classified as chronic active | from baseline to month 6 and month 24
  Percent change in number of plaques classified as chronic active from baseline to month 6 and month 24 in the whole cohort, in RMS cohort (global and splitted in RRMS and RMS having reached the SPMS phase) and in PPMS cohort.
decrease of microglial activation as measured by [18F]DPA-714 PET in number of plaques classified as smoldering plaques | from baseline to month 6 and month 24
  Percent change in number of plaques classified as smoldering plaques from baseline to month 6 and month 24 in the whole cohort, in RMS cohort (global and splitted in RRMS and RMS having reached the SPMS phase) and in PPMS cohort.
decrease of microglial activation as measured by [18F]DPA-714 PET in deep grey matter | between baseline to months 6 and 24
  Percent change in extent of 18FDPA714 positive voxels in deep grey matter between baseline to months 6 and 24 in the whole cohort, in RMS cohort (global and splitted in RRMS and RMS having reached the SPMS phase) and in PPMS cohort.
decrease of microglial activation as measured by [18F]DPA-714 PET in cortical grey matter | between baseline to months 6 and 24
  Percent change in extent of 18FDPA714 positive voxels in cortical grey matter between baseline to months 6 and 24 in the whole cohort, in RMS cohort (global and splitted in RRMS and RMS having reached the SPMS phase) and in PPMS cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Stankoff, MD Ph.D, Principal Investigator — Hôpital Saint-Antoine - Service de Neurologie
Locations (1):
- Hôpital Saint-Antoine - Service de Neurologie, Paris, France